CLINICAL TRIAL: NCT06891976
Title: Effect of Acupressure Versus Kinesotape on Low Back Pain in Women Who Use Intrauterine Device
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dana Abd Elaziz Mansour, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005281
Record Dates: First submitted 2025-03-18; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Acupressure; Athletic Tape; Ibuprofen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupressure therapy + Non-steroidal anti-inflammatory drugs (Experimental): Twenty four females will receive acupressure therapy (3 times per week, for 3 weeks), in addition to Non-steroidal anti-inflammatory drugs (25-50mg/daily).
  Interventions: Other: Acupressure therapy; Drug: Non-steroidal anti-inflammatory drugs
- kinesio tape + Non-steroidal anti-inflammatory drugs (Experimental): Twenty four females will receive kinesio tape (3 times per week, for 3 weeks), in addition to Non-steroidal anti-inflammatory drugs (25-50mg/daily).
  Interventions: Other: kinesio tape; Drug: Non-steroidal anti-inflammatory drugs
- Non-steroidal anti-inflammatory drugs (Other): Twenty four females will receive only Non-steroidal anti-inflammatory drugs (25-50mg/daily).
  Interventions: Drug: Non-steroidal anti-inflammatory drugs

INTERVENTIONS:
Other: Acupressure therapy — It will be applied to the first experimental group, three times per week for 3 weeks, with each session lasting 30 minutes. Each woman will receive a brief explanation about acupressure therapy and its effects to ensure her confidence and cooperation. Before starting, participants will be asked to empty their bladder for relaxation and assume a prone position. The therapy involves applying prolonged, slow, firm pressure with both thumbs on five key points (BL20, GV3, GB30, GB34, and BL25), which are commonly used for low back pain. Each point will receive three cycles of one-minute pressure followed by one minute of relaxation.
  Arms: Acupressure therapy + Non-steroidal anti-inflammatory drugs
Other: kinesio tape — It will be applied to the second experimental group, for 3 weeks. The tape, 5cm wide and 0.5mm thick, will be fixed in a standing lumbar flexion position on clean, grease-free skin. Four I-shaped bands, each 0.5mm in width, will be applied. The first 5cm of tape will be carefully placed on the skin without stretching, while the middle portion will be stretched 1-2 inches (50%). Two bands will be applied horizontally, and two more will be placed vertically along the lumbar spine, from the lower iliac crest to the upper twelfth rib. The tape will be rubbed to warm the adhesive, ensuring proper adhesion. It will be replaced every 3 days for 3 weeks.
  Arms: kinesio tape + Non-steroidal anti-inflammatory drugs
Drug: Non-steroidal anti-inflammatory drugs — All the three groups will receive 400mg of Non-steroidal Anti-Inflammatory Drugs (Ibuprofen) once a day on the treatment days two hours before the session.
  Other Names: Ibuprofen

SUMMARY:
The study will be conducted to differentiate between the effect of acupressure and kinesiotape on low back pain in women who use intrauterine device.

DETAILED DESCRIPTION:
Overall, the Egypt Demographic and Health Survey (EDHS) results indicate that 60% of currently married women in Egypt are using contraception. The IUD, pill, and injectable are the most widely used methods: 36% of currently married women interviewed for the Egypt Demographic and Health Survey (EDHS) use the IUD, 12% rely on the pill, and 7% utilize injectable.

IUD insertion possess numerous complications which includes low back pain, cervical problems, syncope, bradycardia, convulsions, perforation, expulsion, frequent bleeding , all affecting the quality of life of women.

Analgesia has been used by many patients for relieving their low back pain symptoms. Unfortunately, despite of its fast relieving effects, analgesics can cause side effects as heartburn, indigestion, nausea, vomiting, constipation, diarrhea, headaches, dizziness, drowsiness, stomach ulcers and liver damage. This draws the necessity to consider the use of physical therapy modalities for the treatment of low back pain like active exercises, various elecyrotherapy modalities with the emphasis on the use of acupressure and Kinesotape.

Numerous studies have addressed the effect of acupressure on LBP. A previous study showed that acupressure could reduce postpartum LBP intensity. Also, it was reported that applying pressure on specific acupoints reduced LBP among nurses.

Also, previous studies have shown that KT improves blood and lymph circulation, mitigates pain, adjusts joints, and relives muscle tension. Previous research examined the effects of Kinesiotaping on LBP associated with pregnancy and showed that the intensity of LBP was lower in the group of the Kinesiotape and paracetamol than in the group that took paracetamol alone.

Till now there is no previous study differentiate between the effect of kinesiotape and acupressure in the management of low back pain in women with intrauterine device. So, the study will be conducted to determine which of them is more effective on relieving intrauterine device related low back pain which will be of valuable benefits and increased body of knowledge of physical therapists in scientific field.

ELIGIBILITY:
Inclusion Criteria:

* Females suffer from low back pain resulted from intrauterine device use, they are referred by the gynecologist.
* Their pain level will be> 4 on the visual analogue scale (VAS).
* Their ages will be ranged from 25 to 30 years.
* Their BMI will be less than 30 kg /m2
* Women diagnosed with low back pain upon recent insertion of intrauterine device (within a year)
* All patients will be clinically and medically stable when attending the study.

Exclusion Criteria:

* Current pelvic infection, usually pelvic inflammatory disease (PID), mucopurulent cervicitis with a suspected STI, pelvic tuberculosis, septic abortion, or puerperal endometritis or sepsis within the past 3 months
* Unexplained vaginal bleeding
* Patients having skin disease or known allergy to kinesio tape
* Having LBP due to trauma, spondylolisthesis, ankylosing spondylitis, fibromyalgia, diabetes mellitus or due to any gynecological problems that may cause LBP like polycystic ovarian syndrome (PCO), endometriosis, adenomyosis, cervicitis, uterine prolapse etc.

Ages: 25 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-03-25 (Estimated); Primary Completion 2025-05-10 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of pain intensity | 3 weeks
  The visual analog scale (VAS) will be used to assess pain intensity for all participating females in the three groups before and after the study program. It is a horizontal line whose length is 10 cm; its left end (zero) indicates no pain, while its right end (ten) reveals the worst imaginable pain. Each female will be asked to mark a point on the line between the extreme that is related to her pain intensity level.
Assessment of pain pressure threshold | 3 weeks
  A pressure algometer will be used to measure pressure pain thresholds (PPT) for all participants in the three groups before and after the study. PPTs will be assessed at specific marked points on the body. All participants will be instructed to take non-steroidal anti-inflammatory drugs at least 4 hours before the procedure. Two measurements will be taken for the dominant forearm extensor muscle to ensure proper understanding, with a third if needed. Alcohol will clean the evaluation areas. A 1-cm² pressure probe will be used to record PPTs at five marked sites on the lumbar region (L1-S2), with three measurements per site and a 60-second interval between tests. The patient will be in a lateral decubitus position, reporting pain onset, and the mean value will be recorded.

SECONDARY OUTCOMES:
Assessment of functional disability | 3 weeks
  The Arabic version of the Oswestry Disability Index (ODI) will be used to assess functional disability in females in all three groups before and after the study. The ODI consists of ten sections, each with six response options describing functional impairments in daily activities. Scores range from 0 to 5, with the highest score taken if multiple boxes are marked. The total score is calculated by dividing the sum of the scores by the total possible score, multiplied by 100 to get a percentage. If a section is missed, the score is adjusted accordingly. A low score indicates low disability, while a high score indicates a higher degree of disability.

CONTACTS AND LOCATIONS:
Overall Officials: Hala Mohamed Hanfy Omaera, PhD, Study Chair — Professor, Cairo university; Hossam El Deen Kamel, PhD, Study Director — Professor, Al-Azhar university
Locations (1):
- Kasr Al Ainy Hospital, Giza, Egypt